CLINICAL TRIAL: NCT03981783
Title: Comprehensive Health Informatics Engagement Framework for Pulmonary Rehab
Brief Title: Informatics Framework for Pulmonary Rehabilitation
Acronym: CHIEF-PR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph Finkelstein, Chief Research Informatics Officer, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 18-1637; R61HL143317-01 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: COPD
Keywords: COPD; Pulmonary Rehabilitation; Telerehabilitation; Clinical Decision Support; Adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Comprehensive Health Informatics Engagement Framework for Pulmonary Rehabilitation (CHIEF-PR) will facilitate PR referrals, initial assessments, completion rates, and PR maintenance using multi-pronged approach at the healthcare, provider and patient levels that addresses current barriers for PR uptake and completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best available care (BAC) (Active Comparator)
  Interventions: Behavioral: Best available care (BAC)
- Telerehabilitation (TH) (Experimental)
  Interventions: Behavioral: Telerehabilitation (TH)

INTERVENTIONS:
Behavioral: Best available care (BAC) — Eligible patients are assigned to a standard pulmonary rehabilitation program
  Arms: Best available care (BAC)
Behavioral: Telerehabilitation (TH) — Eligible patients are assigned to a pulmonary telerehabilitation program
  Arms: Telerehabilitation (TH)

SUMMARY:
Previous studies clearly established clinical benefits of pulmonary rehabilitation in patients with chronic obstructive pulmonary disease however uptake and completion rate of pulmonary rehabilitation programs by these patients is limited by multiple barriers. The goal of this project to systematically evaluate impact of Comprehensive Health Informatics Engagement Framework for Pulmonary Rehabilitation (CHIEF-PR) in a randomized controlled trial. The main hypothesis is that CHIEF-PR will result in significantly higher rates of completion of a comprehensive pulmonary rehabilitation program.

DETAILED DESCRIPTION:
Previous studies clearly established clinical benefits of pulmonary rehabilitation in patients with chronic obstructive pulmonary disease (COPD) however uptake and completion rate of pulmonary rehabilitation (PR) programs by these patients is limited by multiple barriers. The study team developed a Comprehensive Health Informatics Engagement Framework for Pulmonary Rehabilitation which facilitates patient referral and promotes adherence with pulmonary rehabilitation program using innovative multi-pronged approach. It includes computer-mediated patient counseling to increase patient motivation in joining PR program followed by ongoing home-based support of PR by a telerehabilitation system that monitors patients' progress and allows remote oversight by clinical PR team. The goal of this project is to systematically evaluate impact of Comprehensive Health Informatics Engagement Framework for Pulmonary Rehabilitation (CHIEF-PR) in a randomized controlled trial. The study team's main hypothesis is that CHIEF-PR will result in significantly higher rates of completion of a comprehensive pulmonary rehabilitation program. The study team will enroll 120 COPD patients within 4 weeks of acute exacerbation of COPD into a randomized controlled trial and follow them for 12 months. Patients will be randomly assigned to intervention (CHIEF-PR) and control (best available standard of care) groups. Primary outcome will be completion rate of a comprehensive 3-month PR program. Secondary outcomes will include relevant clinical and patient-reported parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older at the time of randomization;
* Have a physician diagnosis of COPD
* Have moderate to severe COPD according to GOLD classification (Stages II - III)
* Understand spoken English or Spanish
* Urgent care event due to COPD within 4 weeks of enrollment
* Have no other member of the household enrolled in the study

Exclusion Criteria:

* Evidence that the patient may move from the study area before the completion of the study
* Impaired cognitive status as indicated by MMSE<24
* Presence of any health condition, that would preclude participation (e.g., psychiatric diagnosis, unstable cardiovascular condition or physical disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who completed the program | 3 months
  Percent of eligible COPD patients who completed a comprehensive 3-month PR program to assess adherence with pulmonary rehabilitation

SECONDARY OUTCOMES:
6 minute walking distance | 12 months
  The distance covered over a time of 6 minutes
Chronic Respiratory Disease Questionnaire (CRDQ) | 12 months
  Disease-specific quality of life scaled on a 7-point modified Likert Scale from 1 to 7. The total scale ranges from 20 to 140 with higher scores indicate better health-related quality of life.
Short Form-36 (SF-36) | 12 months
  General quality of life - consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
COPD self-efficacy Scale (CSES) | 12 months
  COPD Self-efficacy Scale is a 34 item scale, each item is scored on a 5-point likert scale from 1 to 5. Total scale range from 34 to 170, with higher score indicating lower confidence in managing and controlling dyspnea
Shortness of Breath Questionnaire | 12 months
  Respiratory symptoms assessed by the shortness of breath questionnaire. 21 items scored on a 6 point scale from 0 to 5, with total scale from 0 to 120. Higher score indicates more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Finkelstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Background] Bedra M, McNabney M, Stiassny D, Nicholas J, Finkelstein J. Defining patient-centered characteristics of a telerehabilitation system for patients with COPD. Stud Health Technol Inform. 2013;190:24-6. PMID 23823363
- [Background] Gibbons MC, Wilson RF, Samal L, Lehman CU, Dickersin K, Lehmann HP, Aboumatar H, Finkelstein J, Shelton E, Sharma R, Bass EB. Impact of consumer health informatics applications. Evid Rep Technol Assess (Full Rep). 2009 Oct;(188):1-546. PMID 20629477
- [Background] Jeong IC, Finkelstein J. Remotely controlled biking is associated with improved adherence to prescribed cycling speed. Technol Health Care. 2015;23 Suppl 2:S543-9. doi: 10.3233/THC-150992. PMID 26410522
- [Background] Finkelstein J, Knight A, Marinopoulos S, Gibbons MC, Berger Z, Aboumatar H, Wilson RF, Lau BD, Sharma R, Bass EB. Enabling patient-centered care through health information technology. Evid Rep Technol Assess (Full Rep). 2012 Jun;(206):1-1531. PMID 24422882
- [Background] Finkelstein J, Cha E, Scharf SM. Chronic obstructive pulmonary disease as an independent risk factor for cardiovascular morbidity. Int J Chron Obstruct Pulmon Dis. 2009;4:337-49. doi: 10.2147/copd.s6400. Epub 2009 Sep 24. PMID 19802349
- [Background] Gibbons MC, Wilson RF, Samal L, Lehmann CU, Dickersin K, Lehmann HP, Aboumatar H, Finkelstein J, Shelton E, Sharma R, Bass EB. Consumer health informatics: results of a systematic evidence review and evidence based recommendations. Transl Behav Med. 2011 Mar;1(1):72-82. doi: 10.1007/s13142-011-0016-4. PMID 24073033
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633